CLINICAL TRIAL: NCT06165900
Title: A Multicenter, Randomized Trial of Stereotactic Radiotherapy Combined With Adebrelimab and TCb (Nab-paclitaxel + Carboplatin) Versus Adebrelimab Combined With TCb (Nab-paclitaxel + Carboplatin) in Neoadjuvant Treatment of Triple-negative Breast Cancer
Brief Title: Stereotactic Radiotherapy Combined With Adebrelimab and TCb (Nab-paclitaxel + Carboplatin) in Neoadjuvant Treatment of TNBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Clinical Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUKDEN 08
Record Dates: First submitted 2023-10-06; First posted 2023-12-12 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Stereotactic Radiotherapy; Immunotherapy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; 130-nm albumin-bound paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adebrelimab plus stereotactic radiotherapy and chemotherapy (Experimental)
  Interventions: Drug: adebrelimab plus stereotactic radiotherapy followed by adebrelimab plus chemotherapy (nab-paclitaxel + carboplatin)
- adebrelimab plus nab-paclitaxel + carboplatin (Active Comparator)
  Interventions: Drug: adebrelimab plus chemotherapy (nab-paclitaxel + carboplatin)

INTERVENTIONS:
Drug: adebrelimab plus stereotactic radiotherapy followed by adebrelimab plus chemotherapy (nab-paclitaxel + carboplatin) — Adebrelimab plus radiotherapy phase: radiotherapy was started on the day of the second cycle of adebrelimab administration every other day for 3 fractions; Adebrelimab plus chemotherapy phase: starting within 3-5 weeks after completion of radiotherapy, every 3 weeks for 6 cycles.
  Arms: adebrelimab plus stereotactic radiotherapy and chemotherapy
Drug: adebrelimab plus chemotherapy (nab-paclitaxel + carboplatin) — adebrelimab plus chemotherapy (nab-paclitaxel + carboplatin)
  Arms: adebrelimab plus nab-paclitaxel + carboplatin

SUMMARY:
This study was an open-label, multicenter, randomized study. It is planned to include 136 patients with stage II-III triple negative breast cancer. Eligible subjects will be randomized to receive either the experimental arm: adebrelimab plus stereotactic radiotherapy followed by adebrelimab plus chemotherapy (nab-paclitaxel + carboplatin) or the control arm: adebrelimab plus nab-paclitaxel + carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve breast cancer female patients aged ≥ 18 years and ≤ 75 years;
* Histopathologically confirmed early or locally advanced triple-negative invasive breast cancer according to the latest ASCO/CAP guidelines, meeting the following conditions: (1) pathological type is triple-negative, specifically: ER negative: IHC < 1%, PR negative: IHC < 1%, HER2 negative: IHC 0/1 + or IHC2 + but ISH negative;
* Clinical stage II-III invasive breast cancer with measurable lesions according to RECIST 1.1;
* ECOG score 0-1;
* Able to tolerate preoperative and postoperative adjuvant radiotherapy after assessment by a radiologist;
* Appropriate level of organ function
* Patients voluntarily participate in and sign the informed consent form, are expected to have good compliance and cooperate with the study according to the requirements of the protocol.

Exclusion Criteria:

* Patients with metastatic breast cancer or bilateral breast cancer;
* Patients with inflammatory breast cancer or occult breast cancer;
* Patients received any anti-tumor therapy within 12 months before signing the informed consent form, including chemotherapy, targeted therapy, radiotherapy, endocrine therapy, immunotherapy, biological therapy or tumor embolization;
* Patients previously received PD-1/PD-L1 antibody, CTLA-4 antibody, or other treatments against PD-1/PD-L1 inhibitors;
* Female patients who are pregnant and lactating, female patients who are fertile and have a positive baseline pregnancy test, or female patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial.
* Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia, and the subject has a known history of psychotropic drug abuse, alcoholism ;
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); positive hepatitis B surface antigen (HBsAg) test, or positive hepatitis B core antibody (HBcAb) test followed by positive HBV-DNA test (HBV-DNA test was performed only in patients with negative HBsAg test and positive HBcAb test); positive hepatitis C virus (HCV) antibody test followed by positive HCV-RNA test (HCV-RNA test was performed only in patients with positive HCV antibody test)
* Any other condition that, in the opinion of the investigator, would make the patient inappropriate for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
tpCR | 6 months
  total pathologic complete response

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No